CLINICAL TRIAL: NCT00122031
Title: Deep Brain Stimulation for Treatment-Refractory Major Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Thomas E. Schlaepfer, MD, Professor of Psychiatry and Psychotherapy, University Hospital, Bonn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSG-04-006
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Depression
Keywords: Major Depression; Treatment Refractory Major Depression
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DBS (Experimental)
  Interventions: Device: Deep Brain Stimulation with Medtronic Activa Neurostimulator

INTERVENTIONS:
Device: Deep Brain Stimulation with Medtronic Activa Neurostimulator — Deep brain stimulation (DBS) at 130 Hz
  Other Names: Activa Neurostimulator

SUMMARY:
This study will investigate the use of deep brain stimulation (DBS) to reduce symptom severity and enhance the quality of life for patients with treatment-refractory major depression.

DETAILED DESCRIPTION:
Despite advances in pharmacotherapy and psychotherapy for major depression, a substantial number of patients fail to improve significantly even after years of conventional and experimental interventions. Bilateral deep brain stimulation (DBS) to the region of the anterior capsule/ventral striatum is an adjustable and reversible procedure that may be a more effective treatment for patients with major depression. This study will determine the effectiveness, safety, and tolerability of DBS in patients with treatment-refractory major depression.

ELIGIBILITY:
Inclusion Criteria:

* Major depression (MD), severe, unipolar type
* German mother tongue
* Hamilton Depression Rating Scale (HDRS24) score of > 20
* Global Assessment of Function (GAF) score of < 45
* At least 4 episodes of MD or chronic episode > 2 years
* > 5 years after first episode of MD
* Failure to respond to *adequate trials (>5 weeks at the maximum recommended or tolerated dose) of primary antidepressants from at least 3 different classes;

  * adequate trials (>3 weeks at the usually recommended or maximum tolerated dose) of augmentation/combination of a primary antidepressant using at least 2 different augmenting/combination agents (lithium, T3, stimulants, neuroleptics, anticonvulsants, buspirone, or a second primary antidepressant); *an adequate trial of electroconvulsive therapy [ECT] (>6 bilateral treatments) and; *an adequate trial of individual psychotherapy (>20 sessions with an experienced psychotherapist).
* Able to give written informed consent
* No medical comorbidity
* Drug free or on stable drug regimen at least 6 weeks before study entry

Exclusion Criteria:

* Current or past nonaffective psychotic disorder
* Any current clinically significant neurological disorder or medical illness affecting brain function, other than motor tics or Gilles de la Tourette syndrome
* Any clinically significant abnormality on preoperative magnetic resonance imaging (MRI)
* Any surgical contraindications to undergoing DBS
* Current or unstably remitted substance abuse (aside from nicotine)
* Pregnancy and women of childbearing age not using effective contraception
* History of severe personality disorder

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-07; Primary Completion 2009-04 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) | analyzed at 12 and 24 month after stimulation onset

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | analyzed at 12 and 24 month after stimulation onset

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Schlaepfer, MD, Principal Investigator — University of Bonn; Volker Sturm, MD, Study Director — University of Cologne
Locations (1):
- Department of Psychiatry and Psychotherapy, University of Bonn, Bonn, Germany

REFERENCES:
- [Background] Cohen MX, Axmacher N, Lenartz D, Elger CE, Sturm V, Schlaepfer TE. Good vibrations: cross-frequency coupling in the human nucleus accumbens during reward processing. J Cogn Neurosci. 2009 May;21(5):875-89. doi: 10.1162/jocn.2009.21062. PMID 18702577
- [Background] Lieb K, Schlaepfer TE. Deep-brain stimulation for Parkinson's disease. N Engl J Med. 2006 Nov 23;355(21):2256; author reply 2256. doi: 10.1056/NEJMc062545. No abstract available. PMID 17124028
- [Background] Kosel M, Sturm V, Frick C, Lenartz D, Zeidler G, Brodesser D, Schlaepfer TE. Mood improvement after deep brain stimulation of the internal globus pallidus for tardive dyskinesia in a patient suffering from major depression. J Psychiatr Res. 2007 Nov;41(9):801-3. doi: 10.1016/j.jpsychires.2006.07.010. Epub 2006 Sep 8. PMID 16962613
- [Result] Schlaepfer TE, Cohen MX, Frick C, Kosel M, Brodesser D, Axmacher N, Joe AY, Kreft M, Lenartz D, Sturm V. Deep brain stimulation to reward circuitry alleviates anhedonia in refractory major depression. Neuropsychopharmacology. 2008 Jan;33(2):368-77. doi: 10.1038/sj.npp.1301408. Epub 2007 Apr 11. PMID 17429407
- [Result] Bewernick BH, Hurlemann R, Matusch A, Kayser S, Grubert C, Hadrysiewicz B, Axmacher N, Lemke M, Cooper-Mahkorn D, Cohen MX, Brockmann H, Lenartz D, Sturm V, Schlaepfer TE. Nucleus accumbens deep brain stimulation decreases ratings of depression and anxiety in treatment-resistant depression. Biol Psychiatry. 2010 Jan 15;67(2):110-6. doi: 10.1016/j.biopsych.2009.09.013. PMID 19914605
- [Result] Bewernick BH, Kayser S, Sturm V, Schlaepfer TE. Long-term effects of nucleus accumbens deep brain stimulation in treatment-resistant depression: evidence for sustained efficacy. Neuropsychopharmacology. 2012 Aug;37(9):1975-85. doi: 10.1038/npp.2012.44. Epub 2012 Apr 4. PMID 22473055
- [Derived] Grubert C, Hurlemann R, Bewernick BH, Kayser S, Hadrysiewicz B, Axmacher N, Sturm V, Schlaepfer TE. Neuropsychological safety of nucleus accumbens deep brain stimulation for major depression: effects of 12-month stimulation. World J Biol Psychiatry. 2011 Oct;12(7):516-27. doi: 10.3109/15622975.2011.583940. Epub 2011 Jul 8. PMID 21736514